CLINICAL TRIAL: NCT00429377
Title: Phase 3 Study of Tacrolimus(FK506)for Lupus Nephritis: A Placebo Controlled, Double-Blind Multicenter, Comparative Study
Brief Title: Phase 3 Study of Tacrolimus (FK506) for Lupus Nephritis: A Placebo Controlled, Double-Blind Multicenter, Comparative Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 506-LN02
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Last update posted 2007-01-31 (Estimated); Status verified 2007-01

CONDITIONS: Lupus Nephritis
Keywords: tacrolimus; FK506; lupus nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Tacrolimus

INTERVENTIONS:
Drug: tacrolimus

SUMMARY:
This study consists of a 28-week placebo-controlled double-blind inter-group efficacy study in steroid refractory Lupus Nephritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Steroid refractory lupus nephritis

  * more than 10mg of steroid failed to control disease activity
  * patients who failed to reduce the amount of steroid
  * patients who couldn't increase the amount of steroid due to side effects

Exclusion Criteria:

* Patients who started the immunosuppressant therapy or increased the amount of immunosuppressant within 12 weeks prior to test drug administration
* Patients who received cyclophosphamide puls within 24 weeks prior to test drug administration
* CNS( Central Nerve System) Lupus patients
* hepatic failure patients
* Serum creatinine ≧1.5mg/dL

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64
Dates: Start 2003-06

PRIMARY OUTCOMES:
Change of Lupus Nephritis - Disease Activity Index total score

SECONDARY OUTCOMES:
proteinuria, RBC-urine, serum creatinine, anti ds-DNA antibody, complement (C3)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chubu Region
  - Hokkaido Region
  - Hokuriku Region
  - Kansai Region
  - Kanto Region
  - Shikoku Region
  - Tohoku Region